CLINICAL TRIAL: NCT00470483
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel Group, fMRI and PET Study Comparing Emotional Challenge-induced Regional Cerebral Blood Flow Changes Before and After 8 Weeks of Treatment With Placebo and Paroxetine in Subjects With Social Anxiety Disorder
Brief Title: A Study To Compare Emotional Changes In Subjects With Social Anxiety Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMT106386
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Social Phobia
Keywords: PET; Social Anxiety Disorder; fRMI
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- arm 1 (Active Comparator): Paroxetine treatment during 8 weeks
  Interventions: Drug: Paroxetine treatment during 8 weeks
- arm 2 (Placebo Comparator): Placebo treatment during 8 weeks
  Interventions: Drug: Placebo treatment during 8 weeks

INTERVENTIONS:
Drug: Placebo treatment during 8 weeks — comparator
  Arms: arm 2
Drug: Paroxetine treatment during 8 weeks — treatment drug
  Other Names: Placebo treatment during 8 weeks
  Arms: arm 1

SUMMARY:
To compare by neuroimaging techniques the way Social Anxiety patients respond to public speaking before and after a drug administration

ELIGIBILITY:
Inclusion criteria:

* Outpatient with Social Anxiety Disorder
* The subject is healthy
* Willing to restrict alcohol intake
* Capable of giving informed consent

Exclusion criteria:

* Subjects with depression or any other psychiatric condition
* Subjects positive for HIV or hepatitis
* Subjects taking drugs or other medication
* Pregnant or becoming pregnant during the study
* Subjects who have donated blood
* Subjects who are left-handed
* Subjects with claustrophobia
* Subjects with an electronic device or ferromagnetic metal foreign body

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-01-22 (Actual); Primary Completion 2009-01-07 (Actual); Study Completion 2009-01-07 (Actual)

PRIMARY OUTCOMES:
fMRI BOLD response in the amygdala and insula elicited by the Matching Emotional Face paradigm at baseline and after 8 weeks of treatment. State-anxiety inventory (STAI-S) after the Public Speaking challenge (only patients). | baseline and after 8 weeks

SECONDARY OUTCOMES:
fMRI BOLD response in selected neuroanatomical ROI elicited by the by Resting State and by other exploratory paradigms at baseline (all subjects) and after 8 weeks of treatment with paroxetine compared to placebo (only patients). | baseline and after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study TMT106386 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/TMT106386?search=study&search_terms=TMT106386#rs
- Available data/document: Informed Consent Form: TMT106386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TMT106386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TMT106386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: TMT106386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TMT106386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TMT106386 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register